CLINICAL TRIAL: NCT04317404
Title: Identifying Variables Associated With Steroid-Induced Hyperglycemia Following Intra-articular Knee Injections Among Diabetic Patients
Brief Title: Knee Steroid Injection and Blood Sugar Signatur
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Reed Williams, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 2019-1202
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Diabetes; Knee Osteoarthritis
MeSH Terms: conditions — Diabetes Mellitus; Osteoarthritis, Knee | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Diabetic with Knee Osteoarthritis: HbA1c between 6.5% - 12.0% in the 3 months prior to Visit 1
  Interventions: Drug: 40 mg Triamcinolone acetonide
- Pre-diabetic with Knee Osteoarthritis: HbA1c between 5.6% - 6.4% in the 3 months prior to Visit 1
  Interventions: Drug: 40 mg Triamcinolone acetonide
- Non-diabetic with Knee Osteoarthritis: HbA1c < 5.6% in the 3 months prior to Visit 1
  Interventions: Drug: 40 mg Triamcinolone acetonide

INTERVENTIONS:
Drug: 40 mg Triamcinolone acetonide — Unilateral knee steroid injection

SUMMARY:
A prospective, observational study assessing the relationship between HbA1c level and the post-injection blood glucose signature. Participants will be non-diabetic, pre-diabetic, non-insulin dependent and insulin dependent type 2 diabetic patients who will be receiving a knee steroid injection. All of them will be consented a week prior to the injection, when the CGM sensor will be applied to the back of the upper arm. This will be removed a week after the injection. KOOS survey as well as VAS will be administered. Adverse events (e.g., change in medication or hospitalization) will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the Parkland Outpatient Clinic
* Indication for unilateral knee joint steroid injection for the treatment of knee joint osteoarthritis

Exclusion Criteria:

* Less than 18 years old
* HbA1c > 12.0%
* steroid exposure in the 3 months prior to Visit 1
* 3 or more steroid injections in the preceding 12 months
* known contraindication to steroid injection (adverse reaction or allergy, active infection, INR > 3.0)
* lack of improvement with prior knee steroid injection
* change in diabetic medication regimen in the last 1 month
* significant change in diet within the last 1 month
* current use of aspirin
* allergy to adhesive
* planned MRI, XR, or CT during the 2-week study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Knee joint osteoarthritis requiring knee joint steroid injection
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Post-injection glucose levels | 1 week
  Blood glucose levels after injection of steroid to the knee

SECONDARY OUTCOMES:
Post-injection adverse events | 1 week
  Adverse events after injection of steroid to the knee
KOOS Knee survey | 2 weeks
  KOOS Knee survey administered before and after steroid injection to the knee

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No